CLINICAL TRIAL: NCT04537052
Title: A New Method for Treatment of Deep Venous Insufficiency: Early Results of Vein Restoration Treatment(VRT) Erdinç EROĞLU
Brief Title: A New Method for Treatment of Deep Venous Insufficiency: Early Results of Vein Restoration Treatment(VRT)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Erdinç Eroğlu, Principal Investigator, Kahramanmaras Sutcu Imam University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-2020/01
Record Dates: First submitted 2020-06-01; First posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Primary Varicose Veins
Keywords: Deep venous insufficiency,

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Onl Femoral vein (Experimental): Ultrasound-guided controlled injection begins, and the venous diameter and gap between valves are reduced
  Interventions: Procedure: Ven Restoration Therapy

INTERVENTIONS:
Procedure: Ven Restoration Therapy — This is a novel and promising method, applied percutaneously, in the treatment of deep venous insufficiency . In this method, developed based on the effects of compression garments, a polymer consisting of cyanoacrylate and hyaluronic acid is injected, with ultrasound-guidance, percutaneously around the femoral vein. In this way, the diameter of the vein is reduced, and function is restored to the inadequately functioning valve. The procedure is also called percutaneous valvuloplasty. The underlying idea in the development of this product was that hyaluronic acid might cause an increase in connective tissue, while cyanoacrylate could serve as an exoskeleton by forming heavy tissue.

SUMMARY:
To present the 9. months clinical results of percutaneous Ven Restoration Therapy (VRT), a new method in the treatment of primary femoral vein insufficiency.Twenty four patients diagnosed with isolated primary femoral vein insufficiency between January 2020 and December 2020 were included in the study. Before the procedure, junctional femoral vein diameters and reflux times were measured. CEAP classification and Venous clinical severity scores (VCSS) were recorded. Chronic Venous Insufficiency Questionnaire (CIVIQ-20) were also recorded. Then, VRT was applied percutaneously to the anterior and posterior of the femoral veins of the patients, and the diameter of the femoral vein was narrowed and valve coaptation was achieved. After the procedure, vein diameters and reflux times were measured again. All parameters were reevaluated by calling patients for control at 1.,3., 6. and 9. months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with isolated deep venous insufficiency, without accompanying superficial venous insufficiency,
* volunteering to take part in the study were included

Exclusion Criteria:

* post-thrombotic or congenital deep venous insufficiency
* Venous reflux disease in the GSV diagnosed by clinical symptoms
* Local or systemic infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-09-27 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-01-30 (Estimated)

PRIMARY OUTCOMES:
femoral vein diameters | 9 months
  reduce femoral vein diameter
reflux times | 9 months
  reduce reflux times

IPD SHARING:
Plan to Share IPD: No